CLINICAL TRIAL: NCT04262219
Title: Enhancing Clinician Communication About Sexual Health in Breast Cancer
Brief Title: Clinician Communication About Sexual Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-1068; 1R03CA235238-01 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iShare (Experimental): Participants will be asked to listen to a podcast intervention.
  Interventions: Behavioral: iShare

INTERVENTIONS:
Behavioral: iShare — The iShare intervention consists of a two-episode educational podcast series containing information about breast cancer patients' sexual problems, approaches for addressing sexual concerns, and information about discussing sexual concerns with patients, such as initiating a conversation about sexual health and asking questions to assess sexual concern. Both episodes feature expert guests and relevant discussions or case studies.

SUMMARY:
The objective of this study is to adapt a previously tested brief intervention aimed at enhancing clinicians communication about sexual health (iSHARE) to a mobile web-based platform showcasing a two-part podcast and to assess the feasibility, acceptability, and preliminary effects of the intervention in breast cancer clinicians.

DETAILED DESCRIPTION:
Specific aims are: 1) To assess the feasibility and acceptability of iSHARE in a mobile learning (mLearning) format and 2) To assess the preliminary effects of iSHARE in a mLearning format.

ELIGIBILITY:
Inclusion Criteria:

* Clinician is a medical oncologist or medical oncology advanced practice clinician (Nurse Practitioner, Physician Assistant) who treats breast cancer patients

Exclusion Criteria:

* Clinician has participated in previous pilot study of the intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B Reese, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iShare
Started | 32
Completed | 30
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | iShare
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.28 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
Clinical role [Count of Participants; unit: Participants]
  Oncologist | 22
  Physician Assistant | 3
  Nurse Practitioner | 7
Years of Practice in Oncology [Count of Participants; unit: Participants]
  0-5 Years | 11
  6-10 Years | 7
  11-15 Years | 6
  More than 15 Years | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention Trial - Enrollment
Description: Enrollment will be measured through measures of participant enrollment defined as the percent of eligible candidates approached who enroll in the pilot trial.
Time Frame: Baseline
Population: 33 participants were analyzed because 33 eligible study candidates were approached for enrollment. Of these, 32 participants enrolled.
Measure: Number; unit: percent of eligible study candidates
Arm/Group | iShare
Number analyzed (Participants) | 33
percent of eligible study candidates | 96.97

2. Primary Outcome: Feasibility of the Intervention Trial - Retention
Description: Study retention will defined as percentage of enrolled participants who complete all study surveys.
Time Frame: Baseline up to 1 month
Measure: Number; unit: percentage of participants
Arm/Group | iShare
Number analyzed (Participants) | 32
percentage of participants | 93.75

3. Primary Outcome: Feasibility of the Intervention Trial - Intervention Completion
Description: Intervention completion will defined as percentage of enrolled participants who complete participation in the podcast intervention.
Time Frame: 1 month
Measure: Number; unit: percentage of participants
Arm/Group | iShare
Number analyzed (Participants) | 32
percentage of participants | 93.75

4. Primary Outcome: Acceptability
Description: Acceptability will be measured through the percentage of the sample endorsing 6 primary acceptability items favorably at two time points (1 week and 1 month; satisfaction, informativeness, relevance, ease of listening, likelihood to recommend, likelihood to impact practice).
Time Frame: 1 week up to 1 month
Measure: Number; unit: percentage of participants
Arm/Group | iShare
Number analyzed (Participants) | 30
percentage of participants | 80

5. Primary Outcome: Change in Clinician Knowledge About Sexual Health and Related Communication
Description: Clinician knowledge about sexual health and communication will be measured using a 10-item scale asking about common sexual problems experienced by breast cancer patients and the most effective ways to communicate with patients about these issues. Knowledge scores range from 0 to 10, with higher scores indicating more knowledge.
  Knowledge will be reported as the mean of items answered correctly. Positive mean change scores indicate an increase in knowledge over time.
Time Frame: Baseline up to 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iShare
Number analyzed (Participants) | 30
score on a scale | 1.6 [0.82 to 2.3]

6. Primary Outcome: Change in Clinician Self-Efficacy About Sexual Health Communication
Description: Clinician self-efficacy about sexual health communication will be measured using a 3-item scale asking about confidence in discussing sexual concerns with patients. Mean scores range from 0-10, with higher scores indicating higher self-efficacy. Positive mean change scores indicate an increase in self-efficacy over time.
Time Frame: Baseline up to 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | iShare
Number analyzed (Participants) | 30
units on a scale | 0.76 [0.29 to 1.2]

7. Primary Outcome: Change in Clinician Outcome Expectancies for Sexual Health Communication
Description: Clinician outcome expectancies for sexual health communication will be measured using a 7-item scale asking about expected positive results in discussing sexual concerns with patients. Mean scores range from 0-10, with higher scores indicating better expected outcomes. Positive mean change scores indicate an increase in outcome expectancies over time.
Time Frame: Baseline up to 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | iShare
Number analyzed (Participants) | 30
units on a scale | 0.52 [0.17 to 0.86]

8. Primary Outcome: Change in Clinician Comfort With Communicating About Sexual Health
Description: Clinician comfort with sexual health communication will be measured using a 7-item scale asking about comfort level in discussing sexual concerns with patients. Mean scores range from 0-10, with higher scores indicating a higher level of comfort. Positive mean change scores indicate an increase in comfort level over time.
Time Frame: Baseline up to 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | iShare
Number analyzed (Participants) | 30
units on a scale | 0.80 [0.46 to 1.14]

9. Primary Outcome: Change in Clinician Communication About Sexual Health
Description: Clinician communication about sexual health will be measured using a 3-item scale asking about recent communication practices around sexual health (initiating conversations, offering information, giving referrals). Mean scores range from 1-5, with higher scores indicating higher amounts of communication. Positive mean change scores indicate an increase in communication behaviors over time.
Time Frame: Baseline up to 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | iShare
Number analyzed (Participants) | 30
units on a scale | 0.16 [-0.15 to 0.46]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | iShare
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT04262219/Prot_SAP_000.pdf